## **OFFICIAL TITLE OF THE STUDY:**

EFFECT OF DILUTED THYME HONEY ON DRY MOUTH IN INTENSIVE CARE UNIT PATIENTS EXPOSED TO OXYGEN FLOW THERAPY: A RANDOMİZED CONTROLLED STUDY

**DOCUMENT TYPE: INFORMED CONSENT FORM** 

### **RESEARCHERS:**

- ESRA YAPRAK GÖKTÜRK (MSC)
  ANKARA UNİVERSİTY
  GRADUATE SCHOOL OF HEALT SCİENCES
  - AYTEN DEMİR (PROFESSOR DOCTOR)
    ANKARA UNİVERSİTY
    FACULTY OF NURSING

**DOCUMENT DATE: 30/11/2022** 

ANKARA/TURKEY

# EFFECT OF DILUTED THYME HONEY ON DRY MOUTH IN INTENSIVE CARE UNIT PATIENTS EXPOSED TO OXYGEN FLOW THERAPY: A RANDOMIZED CONTROLLED STUDY

• NCT ID: Not Yet Assigned

#### Correspondance

Esra Yaprak Göktürk (eyk1994.ek@gmail.com) (+905377819714)

#### • Esra Yaprak GÖKTÜRK

Nursing Department Thesis Master's Program, Institute of Health Sciences, Ankara University

eyk1994.ek@gmail.com

Clinical Trials Organization: AnkaraU

**Clinical Trials User: EYGokturk** 

#### • Ayten DEMİR

Faculty of Nursing, Department of Nursing, Ankara University, Ankara Türkiye

aytendemirankara@gmail.com

https://orcid.org/0000-0002-5677-2347

#### • Ethics Statement

To conduct this research, ethics committee approval (number 56786525-050.04.04/737202) dated November 30, 2022, was obtained from the Ankara University Rectorate Ethics Committee. Institutional approval (meeting number 0137) dated September 18, 2022, was obtained from the Ankara Training and Research Hospital, where the research was conducted. This study was completed as a master's

thesis in the Nursing Department program at Ankara University, Institute of Health Sciences.

#### • Data Availability Statement

We have confirmed that the methods used in data analysis are appropriate. They were applied to our data within the study design and context, and the statistical results were applied and interpreted correctly. As a condition of journal submission, we accept responsibility for ensuring that the selection of statistical methods is appropriate and is performed and interpreted correctly. The data and original materials contained in this study can be obtained by contacting Esra Yaprak Göktürk, one of the authors of this study, at eyk1994.ek@gmail.com

#### INFORMED CONSENT FORM

**Study Title:** The effect of diluted thyme honey on dry mouth in intensive care patients receiving nasal oxygen flow therapy: Randomized Controlled Trial

"Dear volunteer, you have been invited to participate in the above-mentioned research. Before you agree to take part in this study, you need to understand the purpose of the study and make your decision freely within the framework of this information. Please read the following information carefully, ask any questions you may have and ask for a clear answer."

The study is of experimental type and will be conducted to examine the effect of thyme honey on dry mouth in intensive care patients who are treated in the Adult General Intensive Care (Emergency Intensive Care Unit) and Emergency Critical Intensive Care Units serving on the 2nd floor of the Ankara Training and Research Hospital Emergency Department Building and receive nasal oxygen flow therapy. It is planned to include 64 patients in the study. The data of the study is planned to be collected between October 1, 2022 and November 30, 2022. The data will be collected using the "Subjective Dry Mouth Assessment Form", "Patient Information Form" and "Patient Follow-up Form". If you agree to participate in the study, you will be asked to complete these data collection forms. It is thought that the application of the data collection forms will take approximately 20-25 minutes. You can fill out these data collection forms in printed form, or if you wish, a link to the online version of the forms will be sent by the researchers to an e-mail (mail) address provided by you and you will be able to fill out the forms online.

"Taking part in this research is entirely voluntary. You can refuse to take part in the study or stop taking part after it has started. Your refusal or withdrawal from this study will not affect the treatment and care you receive from this hospital. No fee will be charged to you or the social security organization you are affiliated with for all applications within the scope of the research. You will not be paid any fee at the end of this research. The results of this research will be used for scientific purposes. If you withdraw from the research or are removed from the research by the researcher, the data about you will not be used. However, once the data is anonymized, you will not be able to withdraw from the research. All information obtained from you will be kept confidential and the confidentiality of your identity information, if any, will be maintained when the research is published."

"I have read (or listened orally) to the text above, which contains the information that should be given to volunteers before starting the study. I have asked my questions to the researchers about the issues that I thought were incomplete and received satisfactory answers. I believe that I have understood all the written and verbal explanations in detail. I was given enough time to decide whether I wanted to participate in the study or not. Under these conditions, I hereby declare that I freely and without any pressure or coercion, agree to the use of my personal information obtained for scientific purposes, and to its presentation and dissemination in accordance with the rules of confidentiality."

| | Tarih | İmza |
|-------------------------------------------------|-------|------|
| Name and surname of the participant: | | |
| Name and surname of the researcher: Esra Yaprak | | |
| GÖKTÜRK | | |

Address: Ankara Üniversitesi Hemşirelik Fakültesi Aktaş Mahallesi Plevne Caddesi. No:5 PK: 06080

Altındağ, Telefon: 0312 319 14 50